CLINICAL TRIAL: NCT02277977
Title: Messung Von Mikrozirkulationsstörungen im Septischen Schock Mit Kontrastmittel- verstärkter Sonographie Evaluation of Impaired Microcirculation During Septic Shock With Contrast Enhanced Ultrasound
Brief Title: Evaluation of Impaired Microcirculation During Septic Shock With Contrast Enhanced Ultrasound
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Principal Investigator, Ingeborg Landerer, Ingeborg Landerer, Clinical Trials Unit, University Hospital Freiburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CUPIDDCH
Record Dates: First submitted 2014-10-27; First posted 2014-10-29 (Estimated); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Sepsis
Keywords: sepsis; septic shock; contrast-enhanced ultrasound; microcirculation
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Contrast enhanced ultrasound (Experimental): Contrast enhanced ultrasound during septic shock
  Interventions: Other: Contrast enhanced ultrasound

INTERVENTIONS:
Other: Contrast enhanced ultrasound — Contrat enhanced ultrasound during septic shock

SUMMARY:
Microcirculatory disorders play a central role in the pathogenesis of sepsis and septic shock. Without adequate therapy that may lead to multi-organ failure and death. Therefore useful therapeutic measures aim to improve the microcirculation, to avoid tissue hypoxia and thus multiple organ failure or death. Clinically, the microcirculation can currently be indirectly evaluated using the diuresis and metabolic parameters (eg, lactate). The aim of the present study is to measure the microcirculation in septic shock by means of contrast-enhanced sonography of the calf muscles. For this purpose, the method is applied to 24 subjects during and after septic shock. It will be investigated in this study whether the microcirculation measurement with ultrasound contrast reflects the severity of the disease. As well as to evaluate whether the use of this diagnostic method could lead to better treatment of the septic shock.

ELIGIBILITY:
Inclusion Criteria:

* septic shock

Exclusion Criteria:

* myocardial infarction

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11 (Estimated); Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Contrast transit time during and after septic shock | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Duerschmied, MD, PHD, Study Director — University of Freiburg